CLINICAL TRIAL: NCT04112576
Title: Physiological Signals, Activity and Posture for Surface Mounted Insertable Cardiac Monitor in Heart Failure Study
Acronym: HAPI-HF
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C2116
Record Dates: First submitted 2019-09-23; First posted 2019-10-02 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure, Systolic; Heart Failure, Diastolic
Keywords: echocardiogram
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFrEF: Participants that are diagnosed with NYHA class II or III heart failure with reduced ejection fraction.
  Interventions: Device: Wearable cardiac monitor
- HFpEF: Participants that are diagnosed with NYHA class II or III heart failure with preserved ejection fraction.
  Interventions: Device: Wearable cardiac monitor

INTERVENTIONS:
Device: Wearable cardiac monitor — Participants will be fitted with a wearable cardiac monitor placed on the skin that measures physiologic signals.

SUMMARY:
To characterize the physiological signals collected from a Wearable Cardiac Monitor (WCM) prototype device in subjects with heart failure and preserved ejection fraction (HFpEF) and compare against signals from subjects with heart failure and reduced ejection fraction (HFrEF).

To evaluate the relationship of physiological signals measured from a wearable cardiac monitor (WCM) prototype device with ECHO measures of systolic and diastolic function

DETAILED DESCRIPTION:
This is a non-randomized, feasibility study that will enroll up to 100 participants clinically diagnosed with HFpEF or HFrEF. Approximately 70% of participants will have HFpEF and 30% will have HFrEF.

There will be one study visit per participant. The study visit includes device placement and data collection during postural changes. Echocardiograms will also be collected throughout the study and at least 30% of participants will undergo a submaximal exercise test. The device will then be removed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA class II or III heart failure defined by symptoms and signs of heart failure
* Documented episode of decompensated heart failure in the past 3 years, which either: a) resulted in a hospital admission (primary diagnosis) or b) was treated in out-patient clinic
* HFrEF defined by documented evidence of EF ≤ 40% OR
* HFpEF defined by documented evidence of:
* EF ≥ 50% and no prior record of EF < 40%
* Evidence of relevant structural heart disease or diastolic dysfunction on echocardiographic as defined in the 2016 ESC guidelines
* Able to understand and willing to provide written informed consent to participate in the trial
* Age 21 years old or greater
* Willing and able to participate in the required testing

Exclusion Criteria:

* Prior hospitalization, CV event or surgery within 6 weeks
* Subject is currently enrolled in another clinical trial (excluding registries) that may interfere with the placement of the study system or include the usage of investigational drugs.
* Patients with Active Implantable Medical Devices
* Known allergy to materials used in the study (adhesive tape, titanium, ECG electrodes)
* Have a prosthetic cardiac valve, previously underwent cardiac valve surgery or have hemodynamically unstable (as judged by local investigator) valvular disease
* Subject is pregnant as indicated by patient record
* Patients with rash or open wound on torso locations where investigational devices will be placed
* Patient deemed as clinically unstable or unsuitable to perform prescribed testing as judged by the local investigator

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are diagnosed with NYHA class II or III heart failure with preserved or reduced ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Physiologic Signal Detection | 12 months
  Characterize differences in cardiac physiology and dynamics between heart failure with preserved ejection fraction and heart failure with reduced ejection fraction patient populations using a wearable cardiac monitor prototype device.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Lam, MD, Principal Investigator — National Heart Center Singapore
Locations (3):
- Northwestern University, Chicago, Illinois, United States
- National Heart Center Singapore, Singapore, Singapore
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No